CLINICAL TRIAL: NCT05539833
Title: A Single-arm, Prospective Clinical Study of KSH01-TCR-T in the Treatment of Refractory/Recurrent Solid Tumors
Brief Title: KSH01-TCRT Solid Tumors
Acronym: KSH01-TCRT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: TCRx Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSH01-TCRT-01
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: TCR-T Cells; Refractory Solid Tumors; Relapsed Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental)
  Interventions: Drug: KSH01 injection

INTERVENTIONS:
Drug: KSH01 injection — TCR-T cell injection

SUMMARY:
1) Safety and efficacy of TCR-T cells in subjects with refractory/relapsed solid tumors. 2) The activation and proliferation of TCR-T cells in the subject, and the survival time.

ELIGIBILITY:
1. Inclusion Criteria:

   * Voluntarily participate in clinical research; fully understand this research and sign informed consent voluntarily; be willing to follow and have the ability to complete all experimental procedures;
   * Male or female, aged 18 to 70 years (inclusive);
   * Subjects with advanced malignant solid tumors confirmed by histology or cytology;

     * Dose escalation phase: subjects who have no standard treatment, or who have failed or relapsed after standard treatment, or who cannot tolerate standard treatment with positive target expression;
     * Dose expansion phase: target-positive subjects who progressed on first-line therapy;
   * HLA-A*02 positive and tumor target positive (target tumor cell staining intensity is divided into 0, 1+, 2+, 3+, >30% of cancer cells express 2+ or 3+ positive positive for the target)
   * All toxicities caused by previous anti-tumor therapy were relieved to grade 0-1 (according to NCI CTCAE version 5.0) or to an acceptable level for inclusion/exclusion criteria. Except for other toxicities such as alopecia and vitiligo that the researchers believe do not pose a safety risk to the subjects;
   * Sufficient organ function (without receiving medical support such as blood transfusion and granulocyte colony-stimulating factor within 14 days before cell reinfusion), defined as follows:
   * Blood system:

     * The neutrophil count (ANC) is not lower than the lower limit of the normal value of the center;
     * White blood cells (WBC) are not lower than the lower limit of the normal value of the center;
     * Platelet count (PLT) is not lower than the lower limit of normal value in our center;
     * Hemoglobin (Hb) not less than 0.8*LLN (lower limit of normal);
   * Liver function:

     * Total bilirubin (TBIL) ≤ 2.0 × upper limit of normal (ULN), Gilbert disease subjects should be ≤ 3 × ULN;
     * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤3×ULN (in the dose expansion phase, subjects with liver metastases or liver cancer can be ≤5×ULN); alkaline phosphatase (ALP) ≤2.5× ULN (subjects with bone metastases, ALP≤5×ULN);
   * Renal function:

     * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 ml/min (Cockcroft-Gault formula: ([140-age]×weight [kg]×[0.85, for women only])/(72×creatinine (mg/dl)));
     * The qualitative urine protein is ≤1+; if the qualitative urine protein is ≥2+, a 24-hour urine protein quantitative examination is required, and if the 24-hour urine protein quantitative <1 g, it is acceptable;
   * Coagulation function:

   Those who did not receive anticoagulation therapy: International normalized ratio (INR), activated partial thromboplastin time (APTT) should be less than or equal to 1.5×ULN; patients with liver metastasis or liver cancer should be less than or equal to 2×ULN;
   * Physical status: Eastern Cooperative Oncology Group (ECOG) score of 0-1;
   * Expected survival period ≥ 12 weeks;
   * According to RECIST 1.1 criteria, there is at least one measurable lesion (dose expansion phase) or an evaluable lesion (dose escalation phase);
   * After assessment, enough PBMC cells can be collected in the subject to prepare autologous TCR-T cells;
   * After evaluation, the prepared autologous TCR-T cells are of sufficient quantity and qualified quality, and can be used for clinical reinfusion of the corresponding dose;
   * Female subjects with fertile potential have a negative blood pregnancy result within 3 days before the cell reinfusion, and are willing to abstain from sex or take medically approved high-efficiency drugs from the time of signing the informed consent to 6 months after the end of the last medication. contraceptive measures (eg, IUDs, condoms);
   * Male subjects are willing to keep abstinence or take medically approved high-efficiency contraceptive measures from the time of signing the informed consent to 6 months after the end of the last medication, and do not donate sperm during this period.
   * All subjects are required to provide tumor tissue specimens that can be used for target analysis, which must be archived specimens or fresh biopsy specimens (bone biopsy specimens are not accepted). Only those with positive target expression can enter the study.
2. Exclusion Criteria:

   * History of severe allergic diseases, severe drug allergy (including unmarketed test drugs), or known allergy to any component of the recommended drugs (including pretreatment drugs) in this program;
   * Those who have received coronary artery reconstruction in the past;
   * Evidence of significant bleeding disorders or other significant bleeding risk:
   * History of intracranial hemorrhage or intraspinal hemorrhage;
   * Tumor lesions invade large blood vessels and have obvious bleeding risk;
   * Thrombosis or embolism occurred within 6 months before cell reinfusion;
   * Clinically significant hemoptysis or tumor hemorrhage occurred within 1 month before cell reinfusion;
   * Anticoagulant therapy for therapeutic purposes (except low molecular weight heparin) has been used within 2 weeks before cell reinfusion;
   * Antiplatelet drugs, such as aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine or cilostazine, were used within 10 days before cell reinfusion azoles, etc.;
   * Received the following treatments or drugs before cell reinfusion:

     * Unhealed wounds, ulcers or fractures within 28 days before cell reinfusion;
     * Inoculated with live attenuated vaccine within 28 days before cell reinfusion;
     * Received nitrosourea or mitomycin C treatment within 6 weeks before cell infusion; received oral fluorouracil treatment 2 weeks before cell infusion or within ●half-lives of the drug (whichever is longer) ;
   * Received corticosteroids within 2 weeks before cell reinfusion, or it is expected that corticosteroid treatment may be required during blood collection, cell collection or cell reinfusion; except for the following cases: short time (≤7 days), dose not higher than 10 mg/d prednisone or equivalent dose of corticosteroids for the prevention or treatment of non-autoimmune conditions; topical, intranasal, intraocular, intraarticular or inhaled corticosteroids;
   * Known leptomeningeal metastases, or uncontrolled or symptomatic central nervous system metastases manifested by clinical symptoms, cerebral edema, spinal cord compression, and/or progressive growth. Subjects with a history of central nervous system metastasis or spinal cord compression are acceptable if they have clearly received treatment and are clinically stable after 8 weeks of discontinuation of anticonvulsants and steroids before cell reinfusion;
   * The existence of any form of primary immunodeficiency;
   * There is any active autoimmune disease, or there is a history of autoimmune disease and relapse is expected (including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, need for bronchial Asthma subjects medically intervened with dilators, except for the following: type 1 diabetes; skin conditions not requiring systemic therapy [eg, vitiligo, psoriasis, alopecia]; hypothyroidism only receiving hormone replacement therapy; childhood Asthma in complete remission without any intervention in adulthood; or others not expected to relapse in the absence of external triggers);
   * Within 6 months before cell reinfusion, the following conditions have occurred: myocardial infarction, severe/unstable angina, clinically significant arrhythmia requiring clinical intervention, cerebrovascular accident/stroke, transient ischemic attack, Subarachnoid hemorrhage, cardiac insufficiency with New York Heart Association (NYHA) class ≥ II;
   * There is currently uncontrollable pleural, pericardial, and ascites effusion;
   * Before cell reinfusion, there are:

     * Congenital Long QT Syndrome
     * Use of a pacemaker
     * Left Ventricular Ejection Fraction (LVEF) < 50%
     * QTcF interval>480 msec (QTcF=QT/(RR^0.33))
     * Cardiac troponin I or T >2.0 ULN
     * Poorly controlled diabetes (fasting blood glucose ≥ 13.3 mM)
     * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
     * Forced expiratory volume in the first second (FEV1) ≤ 60% or those who need supplemental oxygen therapy;
   * Unexplained fever >38.5°C during screening or before cell reinfusion (fever due to tumor can be included in the group as judged by the investigator);
   * Known history of allogeneic organ transplantation;
   * Known history of alcohol abuse, psychotropic substance abuse or drug abuse;
   * Have a clear history of neurological or mental disorders, such as epilepsy, dementia, schizophrenia, etc.;
   * Known to have acquired immunodeficiency syndrome (AIDS);
   * Known severe active viral, bacterial infection, or uncontrolled systemic fungal infection;
   * Positive virological test results (HIV, CMV, HSV, HPV, EBV, syphilis);
   * HBsAg positive or HBcAb positive, and HBV-DNA > 200 IU/mL; HCV-Ab positive, and HCV-RNA higher than the detection limit of the research center;
   * According to the judgment of the investigator, the underlying condition of the subject may increase the risk of receiving the experimental drug treatment, or cause confusion in the interpretation of the toxic reactions and adverse events;
   * Expected to receive any other form of antitumor drug treatment during the study period;
   * Women who are pregnant or breastfeeding;
   * Other investigators deem it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v4.0. | about 2 years
  Subject safety
Changes in overall tumor diameter. | about 2 years
  tumor efficacy

SECONDARY OUTCOMES:
Anti-tumor efficacy | about 5 years
  Subject survival time
Pharmacokinetic profile | about 2 years
  Pharmacokinetic Values of blood test values
Cytokine profile | about 2 years
  Cytokine values of blood test values
Biomarker Features profile | about 2 years
  Biomarker Features values of blood test values
Maximum tolerated dose in subjects. | about 2 years
  Subject safety

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ma, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The first affiliated hospital of Guang Xi medical university, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No